CLINICAL TRIAL: NCT05939622
Title: Prospective Randomized Double Blind Placebo Controlled Study of Efficacy of the Therapy With BRAINMAX® Using Functional Magnetic Resonance Imaging (fMRI) for the Treatment of Patients With Post-COVID Asthenic Syndrome
Brief Title: Efficacy of the Therapy With BRAINMAX® Using fMRI for the Treatment of Patients With Asthenia After COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BRAINMAX_2022
Record Dates: First submitted 2023-07-10; First posted 2023-07-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Asthenia; COVID-19; Functional MRI; Cognitive Impairment
Keywords: Asthenia; COVID-19; Chronic fatigue syndrome; Functional MRI; Cognitive impairment; Brain fog; BRAINMAX
MeSH Terms: conditions — Asthenia; COVID-19; Cognitive Dysfunction; Fatigue Syndrome, Chronic; Mental Fatigue | interventions — 3-(2,2,2-trimethylhydrazine)propionate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fMRI with subsequent injection of active drug (Ethyl methyl hydroxypyridine succinate + Meldonium) (Experimental): Arm 1 (n=15) performed structural and functional MRI and received intramuscularly with the dosage regimen of 5 mL of solution (500 mg of ethyl methyl hydroxypyridine succinate + 500 mg of meldonium) once per day for 10 days
  Interventions: Other: Structural and functional MRI; Drug: Ethyl methyl hydroxypyridine succinate + Meldonium
- fMRI with subsequent injection of placebo (Placebo Comparator): Arm 2 (n=15) performed structural and functional MRI and received Placebo in the same way.
  Interventions: Other: Structural and functional MRI; Drug: Placebo

INTERVENTIONS:
Other: Structural and functional MRI — MRI using a Siemens MAGNETOM Prisma 3T scanner before and after a course of therapy, using resting state fMRI and with cognitive paradigm.
  Other Names: fMRI
Drug: Ethyl methyl hydroxypyridine succinate + Meldonium — Ethyl methyl hydroxypyridine succinate 100.0 mg/mL, meldonium dihydrate - 100.0 mg/mL (Solution for intravenous and intramuscular administration)
  Other Names: BRAINMAX®
  Arms: fMRI with subsequent injection of active drug (Ethyl methyl hydroxypyridine succinate + Meldonium)
Drug: Placebo — Placebo was used in the same way
  Arms: fMRI with subsequent injection of placebo

SUMMARY:
to assess executive network using resting-state fMRI and patterns of brain activation using task fMRI with a cognitive paradigm, against the background of taking the drug in comparison with placebo in patients with post-COVID asthenic syndrome.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, placebo-controlled trial to evaluate the effectiveness of therapy using functional MRI of the brain in the setting of neuroprotective therapy for the treatment of patients with chronic fatigue syndrome after COVID-19. The study included 30 patients matched by sex and age with confirmed coronavirus infection. All patients were examined with MFI-20, MoCa, FAS-10 scales, MRI using a Siemens MAGNETOM Prisma 3T scanner before and after a course of therapy with EMHPS-M or placebo (15 patients each) using resting state fMRI and with cognitive paradigm. First group received intramuscularly with the dosage regimen of 5 mL of solution (500 mg of ethyl methyl hydroxypyridine succinate + 500 mg of meldonium) once per day for 10 days. Second group received Placebo in the same way.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to sign the patient informed consent form for the participation in the clinical study
* Patients of both sexes of 25-50 years of age
* Patient's negative test result for severe acute respiratory syndrome (SARS) -CoV-2 RNA obtained by polymerase chain reaction (PCR) method within 72 hours
* COVID-19 diagnosis documented in the history more than 12 weeks ago*
* Symptoms of Post-COVID-19 syndrome (asthenic state, feeling of energy loss and decreased functioning, intellectual function disorder, attention and memory disorder, emotional lability, reducing stress resistance) which appeared during or after COVID-19, retain for more than 12 weeks and cannot be explained by an alternative diagnosis
* Patients capable of following the requirements of the Clinical Study Protocol
* Negative pregnancy test result (for women with the active childbearing potential)
* MFI-20 scale score is more than 30 at the moment of screening.
* Higher education.
* Lack of decompensated somatic pathology
* Lack of indications of the transferred/current disease of the nervous system

Exclusion Criteria:

* Allergic reactions to the components of the study product
* Taking prohibited drugs/dietary supplements during the previous randomization of the month
* Severe hepatic failure
* Severe renal failure
* Chronic liver and hepatic diseases
* Thyroid diseases
* Anaemia
* Malignant tumour of any localization currently or during 5 years before the inclusion into the study except for completely treated carcinoma in situ
* Autoimmune diseases
* Other chronical diseases which, according to the investigator, can cause asthenia
* Pregnancy or lactation period
* Tuberculosis, cancers or positive reaction to the HIV infection, hepatitis B & C, syphilis according to the history data
* Severe eyesight and/or hearing disorders, serious articulation disorders and/or other deviations able to prevent the patient from adequate cooperation during the study)
* Mental disorders in the history
* Alcohol, drug abuse or drug dependence in the history
* Patients which, according to the investigator, are obviously or probably incapable of understanding and evaluating this study information within the process of the informed consent form signing, including but not limited to with regard to expected risks and possible discomfort
* Other diseases, symptoms or conditions not listed above, which, according to the investigator, are predicaments for the participation in the clinical study
* The presence of contraindications for MRI
* The presence of contraindications for taking the drug

Contraindications for MRI:

* Electronic medical devices in the body (cardiomyostimulator and other)
* Metal elements in the study area (prosthesis, clamp, fragment)
* Invariable behavior of patients
* Inability to remain still during MRI

Prohibited drugs/dietary supplements:

* Ethyl methyl hydroxypyridine succinate and Meldonium (other than the one studied in the study)
* Psychotropic medication
* Drugs containing succinic acid and its salts
* Drugs containing vitamin B6 and /or its derivatives
* Antioxidants, antihypoxic drug and metabolic drugs
* Nootropic drugs

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Changing patterns of brain activation using task fMRI with a cognitive paradigm | From baseline to Visit 2 (day 10)
  Changing patterns of brain activation using task fMRI with a cognitive paradigm, against the background of taking Brainmax in comparison with placebo in patients with post-COVID asthenic syndrome.

SECONDARY OUTCOMES:
Asthenia on a scale Multidimensional Fatigue Inventory (MFI-20) after the completion of the parenteral therapy | From baseline to Visit 2 (day 10)
  MFI-20 has an even proportion of positively and negatively worded items that are rated on a 5-point Likert scale. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue.
  Mean decrease of MFI-20 asthenia scale score after the completion of the parenteral therapy
Fatigue on a Fatigue Assessment Scale (FAS-10) scale after the completion of the parenteral therapy | From baseline to Visit 2 (day 10)
  The FAS is a 10-item general fatigue questionnaire to assess fatigue. Five questions reflect physical fatigue and 5 questions (questions 3 and 6-9) mental fatigue. Subsequently, the total FAS score can be calculated by summing the scores on all questions (recoded scores for questions 4 and 10). The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
  Score dynamics by FAS-10 scale after the completion of the parenteral therapy
Cognitive function on a Montreal Cognitive Assessment (MoCA) scale after the completion of the parenteral therapy | From baseline to Visit 2 (day 10)
  The Montreal Cognitive Assessment (MoCA) is a test used by healthcare providers to evaluate people with memory loss or other symptoms of cognitive decline. Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.
  Score dynamics by MoCA scale after the completion of the parenteral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marine Tanashyan, MD, PhD, Principal Investigator — Federal State Budgetary Research Institution "Research Centre of Neurology"
Locations (1):
- Federal State Budgetary Research Institution "Research Centre of Neurology", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No